CLINICAL TRIAL: NCT04879823
Title: Post-operative Course of Dexamethasone to Reduce Tonsillectomy Morbidity
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: David Chi, MD (Other)
Responsible Party: Sponsor-Investigator, David Chi, MD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY20120036
Record Dates: First submitted 2021-05-04; First posted 2021-05-10 (Actual); Results first posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Adenotonsillectomy; Analgesia; Surgery
Keywords: Pediatric Otolaryngology; Steroid; Placebo; Post-operative pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Dexamethasone; Ibuprofen; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Double blind placebo controlled randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone (Experimental): IV Dexamethasone Sodium Phosphate will be prescribed orally at a dose of 0.5mg/kg with a max dose of 20mg to be taken the morning of days 2, 4, and 6 post-operatively. The Dexamethasone will be mixed by the parents with 5mL of pre-packaged cherry syrup.
  Patients will also receive acetaminophen and ibuprofen. Acetaminophen will be prescribed at 15mg/kg to be taken every 4 hours for the first three days, except when sleeping. Ibuprofen will be prescribed at 10 mg/kg to be taken every 6 hours for the first three post-operative days.
  Patients and parents/caregivers will be asked to complete a pain diary which will be used to determine the level of pain control achieved with this regimen. Families will also be asked daily to check symptoms that were experienced by the child and their child's current comfortable diet. The diary will be completed by post-operative day 14. The diary will be returned via email, mail, or a post-operative appointment at the main hospital.
  Interventions: Drug: Dexamethasone; Drug: Ibuprofen; Drug: Acetaminophen
- Placebo (Placebo Comparator): An equal volume of water will be prescribed to patients (0.5mg/kg) with a max dose of 20mg to be taken the morning of days 2, 4, and 6 post-operatively. The placebo (water) will be mixed by the parents with 5mL of pre-packaged cherry syrup.
  Patients will also receive acetaminophen and ibuprofen. Acetaminophen will be prescribed at 15mg/kg to be taken every 4 hours for the first three days, except when sleeping. Ibuprofen will be prescribed at 10 mg/kg to be taken every 6 hours for the first three post-operative days.
  Patients and parents/caregivers will be asked to complete a pain diary which will be used to determine the level of pain control achieved with this regimen. Families will also be asked daily to check symptoms that were experienced by the child and their child's current comfortable diet. The diary will be completed by post-operative day 14. The diary will be returned via email, mail, or a post-operative appointment at the main hospital.
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen; Drug: Placebo

INTERVENTIONS:
Drug: Dexamethasone — IV Dexamethasone Sodium Phosphate will be prescribed orally at a dose of 0.5mg/kg with a max dose of 20mg to be taken the morning of days 2, 4, and 6 post-operatively. The Dexamethasone will be mixed by the parents with 5mL of pre-packaged cherry syrup
  Arms: Dexamethasone
Drug: Ibuprofen — Ibuprofen will be prescribed at 10 mg/kg to be taken every 6 hours for the first three post-operative days. After the first three days, the subject should take the ibuprofen every 6 hours as needed for pain control. The daily dose of ibuprofen is not to exceed 1200mg or more than 4 individual doses. It will be prescribed in liquid suspension form for ease of use in pediatric populations. Subjects or parents will purchase this medication and dosage will be given to subjects in easy-to-understand language.
Drug: Acetaminophen — Acetaminophen will be prescribed at 15mg/kg to be taken every 4 hours for the first three days, except when sleeping. After the first three days, the subject should take the acetaminophen every 4 hours as needed for pain control. The daily dose of acetaminophen is not to exceed 5 doses in 24 hours. It will be prescribed in liquid suspension form for ease of use in pediatric populations. Subjects or parents will purchase this medication and dosage will be given to subjects in easy-to-understand language.
Drug: Placebo — An equal volume of water will be prescribed to patients (0.5mg/kg) with a max dose of 20mg to be taken the morning of days 2, 4, and 6 post-operatively. The placebo (water) will be mixed by the parents with 5mL of pre-packaged cherry syrup.
  Arms: Placebo

SUMMARY:
The goal of this study is determine if an oral systemic course of steroids is a safe and effective option in lowering pain and complications following adenotonsillectomy in various pediatric age groups. A double blind, placebo-controlled randomized clinical trial of steroids (dexamethasone) versus placebo postoperatively will be performed. Investigators will determine if there is a difference in post-operative pain and complications between groups.

DETAILED DESCRIPTION:
Purpose: To determine if post-operative dexamethasone is a safe and effective option in the reduction of post-operative pain and morbidity following adenotonsillectomy in various pediatric age groups.

Methods: The subject population will be patients between the ages of 3 and 17 who will undergo adenotonsillectomy. The study will consist of two double-blinded arms - patients receiving a course of oral dexamethasone (doses on post-operative days 2, 4, and 6; 0.5 mg/kg; max dose: 20 mg) in addition to standard pain control regimen and patients receiving an oral placebo course in addition to standard pain control regimen. In the diary they will receive, patients or caregivers will record when specific pain medications were taken each day, a symptoms survey, and pain ratings measured by the Wong-Baker FACES Pain Rating Scale. Patients are able to return their diary at a post-operative appointment at CHP Main, through email by scanning the diary or taking pictures with their phone, or through mailing in the survey in a pre-stamped envelope. Demographic information such as age, race, gender, and household income will be extracted from the diary and the electronic medical record. Information such as surgical technique, concurrent operations, post-operative pain prescription (types, weight based dosage, and total days prescribed) will be extracted from the electronic medical record and recorded as well. Outcomes measured will include pain scale rating and rates of complications between the two groups.

Significance: If it can be demonstrated that dexamethasone after adenotonsillectomy can reduce pain, complications, or need for opioid analgesics without appreciable side effects, a strong argument can be made for the addition of this inexpensive medication to routine post-operative adenotonsillectomy care. This would help with limiting the burden of clinical course of tonsillectomy.

The primary and secondary outcome measures were refined prior to analysis. Originally, the primary outcome measure was "average pain burden" defined as "average pain over 14 post-operative days before and after medications." However, study medication was not administered until day 2, and the power analysis was based on a study by Palme et al (2000) that compared mean pain ratings on postoperative days 2-8. Therefore, the primary outcome was revised to "average pain over 2-8 post-operative days before medications." Average pain over 2-8 post-operative after medications was added as a secondary outcome. The original primary outcome combined analysis of pain before and after medication into one measure. However, pain scores were more commonly reported prior to medication than after. Due to missing post-medication scores, it was determined that the analysis would be more appropriately conducted separately for pain scores before and after medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 3 - 17 undergoing adenotonsillectomy meet inclusion criteria

Exclusion Criteria:

* Patients with Down syndrome
* Patients with a history of coagulopathy
* Patients with craniofacial abnormalities other than plagiocephaly or submucous cleft palate (SMCP)
* Caregivers who cannot speak, read, or write in English proficiently
* Patients who take systemic corticosteroids during the enrollment period
* Patients who take opioids during the enrollment period
* Patients who take chronic opioids
* Patients who are pregnant
* Patients with allergy to or contraindication for taking any of the study medications
* Patients who have the inability to communicate
* Patients who have the inability to localize pain
* Patients who have type 1 diabetes
* Patients who have type 2 diabetes

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 222 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-07-11 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Chi, MD, Principal Investigator — Clinical Director, Division of Pediatric Otolaryngology, UPMC Children's Hospital of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Hospital North Surgery Center, Sewickley, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Only co-investigators as listed under the University of Pittsburgh IRB (Institutional Review Board) protocol for this study will have access to all data and analysis. Data will be shared via UPMC-associated OneDrive and will only be shared between these investigators.

REFERENCES:
- [Background] Gerbershagen HJ, Aduckathil S, van Wijck AJ, Peelen LM, Kalkman CJ, Meissner W. Pain intensity on the first day after surgery: a prospective cohort study comparing 179 surgical procedures. Anesthesiology. 2013 Apr;118(4):934-44. doi: 10.1097/ALN.0b013e31828866b3. PMID 23392233
- [Background] Whelan RL, McCoy J, Mirson L, Chi DH. Opioid prescription and postoperative outcomes in pediatric patients. Laryngoscope. 2019 Jun;129(6):1477-1481. doi: 10.1002/lary.27614. Epub 2018 Dec 26. PMID 30585626
- [Background] Borgstrom A, Nerfeldt P, Friberg D. Postoperative pain and bleeding after adenotonsillectomy versus adenotonsillotomy in pediatric obstructive sleep apnea: an RCT. Eur Arch Otorhinolaryngol. 2019 Nov;276(11):3231-3238. doi: 10.1007/s00405-019-05571-w. Epub 2019 Aug 3. PMID 31377901
- [Background] Titirungruang C, Seresirikachorn K, Kasemsuwan P, Hirunwiwatkul P. The use of steroids to reduce complications after tonsillectomy: a systematic review and meta-analysis of randomized controlled studies. Eur Arch Otorhinolaryngol. 2019 Feb;276(2):585-604. doi: 10.1007/s00405-018-5202-2. Epub 2018 Nov 17. PMID 30448929
- [Background] Macassey E, Dawes P, Taylor B, Gray A. The effect of a postoperative course of oral prednisone on postoperative morbidity following childhood tonsillectomy. Otolaryngol Head Neck Surg. 2012 Sep;147(3):551-6. doi: 10.1177/0194599812447776. Epub 2012 May 14. PMID 22585378
- [Background] Redmann AJ, Maksimoski M, Brumbaugh C, Ishman SL. The effect of postoperative steroids on post-tonsillectomy pain and need for postoperative physician contact. Laryngoscope. 2018 Sep;128(9):2187-2192. doi: 10.1002/lary.27167. Epub 2018 Mar 24. PMID 29573428
- [Background] Greenwell AG, Isaiah A, Pereira KD. Recovery After Adenotonsillectomy-Do Steroids Help? Outcomes From a Randomized Controlled Trial. Otolaryngol Head Neck Surg. 2021 Jul;165(1):83-88. doi: 10.1177/0194599820973250. Epub 2020 Nov 24. PMID 33228459
- [Background] Garra G, Singer AJ, Taira BR, Chohan J, Cardoz H, Chisena E, Thode HC Jr. Validation of the Wong-Baker FACES Pain Rating Scale in pediatric emergency department patients. Acad Emerg Med. 2010 Jan;17(1):50-4. doi: 10.1111/j.1553-2712.2009.00620.x. Epub 2009 Dec 9. PMID 20003121
- [Background] Palme CE, Tomasevic P, Pohl DV. Evaluating the effects of oral prednisolone on recovery after tonsillectomy: a prospective, double-blind, randomized trial. Laryngoscope. 2000 Dec;110(12):2000-4. doi: 10.1097/00005537-200012000-00003. PMID 11129008
- [Background] Feinberg AE, Chesney TR, Srikandarajah S, Acuna SA, McLeod RS; Best Practice in Surgery Group. Opioid Use After Discharge in Postoperative Patients: A Systematic Review. Ann Surg. 2018 Jun;267(6):1056-1062. doi: 10.1097/SLA.0000000000002591. PMID 29215370
- [Background] Monitto CL, Hsu A, Gao S, Vozzo PT, Park PS, Roter D, Yenokyan G, White ED, Kattail D, Edgeworth AE, Vasquenza KJ, Atwater SE, Shay JE, George JA, Vickers BA, Kost-Byerly S, Lee BH, Yaster M. Opioid Prescribing for the Treatment of Acute Pain in Children on Hospital Discharge. Anesth Analg. 2017 Dec;125(6):2113-2122. doi: 10.1213/ANE.0000000000002586. PMID 29189368

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexamethasone | Placebo
Started | 110 | 112
Completed | 62 | 73
Not Completed | 48 | 39
Not completed — Physician Decision | 3 | 1
Not completed — Protocol Violation | 2 | 3
Not completed — Lost to Follow-up | 43 | 35

BASELINE CHARACTERISTICS:
Population: Excludes patients withdrawn due to protocol violation and physician decision
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexamethasone | Placebo | Total
Number analyzed (Participants) | 105 | 108 | 213
Age, Continuous [Median (Full Range); unit: years] | 7.1 [3.1 to 17.6] | 6.9 [3.2 to 17.7] | 7.1 [3.1 to 17.7]
Age, Customized [Count of Participants; unit: Participants]
  3-7 years old | 60 | 60 | 120
  8-12 years old | 31 | 31 | 62
  13-17 years old | 14 | 17 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 54 | 102
  Male | 57 | 54 | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 97 | 102 | 199
  Unknown or Not Reported | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 91 | 94 | 185
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 105 | 108 | 213
BMI Percentile at Baseline [Median (Full Range); unit: percentile] | 81.04 [0.07 to 100.00] | 83.77 [1.70 to 99.99] | 83.24 [0.07 to 100.00]

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Over 2-8 Post-operative Days Before Medications
Description: Average pain over 2-8 post-operative days before medications. This is quantified using the validated Wong-Baker FACES pain metric. The scale is from 0 to 10 with 10 being worse outcome. Patients receive a take-home pain diary and for 14 days report their maximum pain both before and after taking each pain medication. The mean of the pain ratings prior to taking pain medications from post-operative days 2-8 will be the primary outcome measure.
Time Frame: 2-8 days post-operatively
Population: Includes only patients who returned their pain diary (completed the study).
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 62 | 73
score on a scale | 4.2 [3.7 to 4.7] | 4.9 [4.4 to 5.4]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Null hypothesis: Average pain scores before medication will not be lower in the dexamethasone group compared with the placebo group; Test type: Superiority; p = 0.03, t-test, 1 sided

2. Secondary Outcome: ED (Emergency Department) or Urgent Care Visits
Description: Number of emergency department or urgent care visits in 30 post-operative days - assessed via the electronic medical record and the take-home pain diary.
Time Frame: 30 days post-operatively
Population: Excludes patients withdrawn due to protocol violations or physician decision.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 105 | 108
Participants
  0 ED or Urgent Care Visits | 97 | 91
  1 ED or Urgent Care Visit | 5 | 14
  2 ED or Urgent Care Visits | 3 | 2
  3 ED or Urgent Care Visits | 0 | 1
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Null hypothesis: There will be no difference in the proportion of patients visiting the emergency department or urgent care (at least 1 time) post-operatively between dexamethasone and placebo groups; Test type: Superiority; p = 0.07, Fisher Exact

3. Secondary Outcome: Average Pain Burden Post-medication
Description: Average pain over 2-8 post-operative days after medications. This is quantified using the validated Wong-Baker FACES pain metric. The scale is from 0 to 10 with 10 being worse outcome. Patients receive a take-home pain diary and for 14 days report their maximum pain both before and after taking each pain medication. The mean of the pain ratings one hour after talking pain medications from post-operative days 2-8 will be a secondary outcome measure.
Time Frame: 2-8 days post-operatively
Population: Includes only patients who returned their pain diary (completed the study). One patient in the placebo group reported no post-medication pain scores.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Dexamethasone | Placebo
Number analyzed (Participants) | 62 | 72
score on a scale | 2.3 [0.0 to 8.0] | 2.2 [0.0 to 7.3]
Statistical Analysis 1: Comparison: Dexamethasone vs Placebo; Null hypothesis: Average pain scores after medication will not be lower in the dexamethasone group compared with the placebo group; Test type: Superiority; p = 0.98, Wilcoxon (Mann-Whitney)

4. Other Pre Specified Outcome: Number of Readmissions
Description: Number of hospitalizations after discharge in 30 days - assessed using the electronic medical record and the take-home pain diary.
Time Frame: 30 days post-operatively
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Frequency of Each Analgesic Used
Description: In the take-home pain diary, patients will place an 'x' on each time block every day that medication was given for each of the three medications. The frequencies will be summed for a total number and averaged within each group to determine the average number of times of each analgesic used.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Duration of Each Analgesic Used
Description: Using the results of the take-home pain diary, the average number of days of use of each analgesic for each group will be calculated. The last day after which there is no subsequent use of analgesic will define the end-point of the duration of use.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Pain Relief Satisfaction
Description: Score assigned by the patient at the end of 14 post-operative days in the take-home pain diary using a 5-point Likert scale of 0 (strongly disagree) to 4 (strongly agree). Patients will respond to the following statement "I am happy with the pain relief I received in the last 14 days" with responses ranging from strongly agree to strongly disagree. The responses will be assigned a numerical value and the average value for all subjects in the group will be reported as the overall pain relief satisfaction. Higher scores indicate a better outcome.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Frequency of Request for Opioid Medication
Description: Number of requests for opioid medication in 14 post-operative days - assessed via the electronic medical record and the take-home pain diary.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Frequency of Post-operative Oropharyngeal Bleed
Description: Number of post-operative oropharyngeal bleeds in 30 post-operative days - assessed via the electronic medical record.
Time Frame: 30 days post-operatively
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Need for Follow-up Appointment
Description: Does the parent/guardian believe his/her child would require a follow-up appointment - assessed using the individual pain diary.
Time Frame: Two months post-operatively
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Household Income
Description: Total household income ranges will be assessed in the take-home pain diary and reported.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Education Level
Description: Using the take-home pain diary, parents/guardians of the patients will identify the highest level of education achieved by anyone in the household.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Side Effects of Medications
Description: Number of side effects assessed daily including bleeding from mouth or throat, anxiety, difficulty breathing, nausea or vomiting, stomach pain/discomfort, fever (100.4F and higher)
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Night-time Awakenings
Description: Number of night-time awakenings reported in 14 days - assessed via the take-home pain diary.
Time Frame: 14 days post-operatively
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Post-operative Nursing Phone Calls
Description: Number of post-operative phone calls to nursing staff, obtained using the electronic medical record up to 30 days post-operatively.
Time Frame: 30 days post-operatively
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Duration of Hospital Admission
Description: Number of days in the hospital after surgery in 30 post-operative days - assessed via the electronic medical record
Time Frame: 30 days post-operatively
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5-9 weeks depending on the date of the follow-up appointment
Description: Number at risk excludes patients withdrawn due to protocol violations or physician decision. These patients were instructed not to administer any study medication. One of these patients had surgery cancelled after consent was obtained.
Arm/Group | Dexamethasone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/108
Serious Adverse Events (participants affected / at risk) | 3/105 | 8/108
Other Adverse Events (participants affected / at risk) | 5/105 | 10/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone (N=105) | Placebo (N=108)
Post-Tonsillectomy Hemorrhage Requiring Operative Intervention (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Post-Tonsillectomy Hemorrhage with Inpatient Admission but Not Requiring Operative Intervention (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Dehydration Requiring Inpatient Admission (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dexamethasone (N=105) | Placebo (N=108)
Post-Tonsillectomy Hemorrhage Requiring Neither Operative Intervention nor Inpatient Admission (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Emergency Department Visit for Post-Operative Pain (General disorders) | 1 (1) | 8 (8)
Emergency Department Visit for Post-Operative Nausea or Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2)
Surgical Site Infection (Infections and infestations) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination due to slow recruitment in older cohorts (8-12 and 13-17-year-olds) leading to small numbers of subjects analyzed in those age groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-26): https://cdn.clinicaltrials.gov/large-docs/23/NCT04879823/Prot_SAP_000.pdf